CLINICAL TRIAL: NCT03008577
Title: The Impact of Ambient Cesarean Room Temperature on Neonatal Morbidity
Brief Title: Hypothermia and the Effect of Ambient Temperature 2
Acronym: HEAT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Parkland Health and Hospital System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU 062016-040
Record Dates: First submitted 2016-12-28; First posted 2017-01-02 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Hypothermia; Neonatal Outcome; Cesarean Section
MeSH Terms: conditions — Hypothermia

ARMS (2):
- Ambient operating room temperature of 67°F (No Intervention): These patients will have an operating room temperature of 67°F for cesarean delivery, the standard of care at our institution.
- Ambient operating room temperature of 75°F (Active Comparator): Intervention: Ambient operating room temperature of 75°F for cesarean delivery, which is closer to World Health Organization recommendations.
  Interventions: Other: Change in ambient operating room temperature

INTERVENTIONS:
Other: Change in ambient operating room temperature
  Arms: Ambient operating room temperature of 75°F

SUMMARY:
Neonatal hypothermia is associated with increased risk of mortality as well as multiple morbidities. The prior HEAT study conducted at our institution showed a difference in neonatal hypothermia with a change in ambient operating room temperature. The investigator's objective is to determine if an increase in ambient operative room temperature decreases the rate of neonatal morbidity. Operating room temperature will be randomized to the current institutional standard of 20°C (67°F) or a temperature of 24°C (75°F), on a weekly basis for a period of 1.2 years.

DETAILED DESCRIPTION:
This is an open, prospective, randomized, single center trial that will address the primary research question: Does an increase in ambient operating room temperature result in a lower rate of composite neonatal morbidities? During the 1.2 year study period, the operating room temperatures on labor and delivery will be adjusted to either the current standard of care with ambient operating room temperature of 20°C (67°F), or the maximum temperature allowable per hospital policy in the current operating rooms, which is 24°C (75°F), as determined by cluster randomization. Composite neonatal morbidities will be recorded including hypoglycemia necessitating treatment; need for respiratory support within the first 24 hours; culture-proven sepsis; and mortality. Association of outcomes with the types of passive and active warming performed will include these morbidities stratified by gestational age as well as maternal outcomes. In addition, an electronic survey will be administered to the operating resident physicians to assess their experience with the study conditions.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women and their neonates undergoing cesarean delivery by the Parkland Hospital Obstetrics Service on the Labor and Delivery unit during the study period.

Exclusion Criteria:

* Exclusion criteria include cases where a cesarean delivery is planned but a precipitous vaginal delivery occurs, intrauterine fetal demise has been diagnosed prior to start of surgery, the neonate is noted to have a major congenital anomaly and resuscitative efforts are not performed ("comfort care only" provided), or a neonatal temperature is not available.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5221 (Actual)
Dates: Start 2016-08; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Neonatal Composite Morbidities | Up to 24 hours following delivery
  Need for respiratory support, Hypoglycemia necessitating treatment, Culture-proven sepsis; Mortality

SECONDARY OUTCOMES:
Maternal Recovery Room Dwell Times after Cesarean | Up to 48h following delivery
Maternal Hypothermia | Up to 24 hours after delivery
  An oral temperature of less than 36.5C

CONTACTS AND LOCATIONS:
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States

REFERENCES:
- [Derived] Ambia AM, Duryea EL, Wyckoff MH, Tao W, McIntire DD, Seasely AR, Moussa M, Leveno KJ. A Randomized Trial of the Effects of Ambient Operating Room Temperature on Neonatal Morbidity. Am J Perinatol. 2024 May;41(S 01):e1553-e1559. doi: 10.1055/a-2053-7242. Epub 2023 Mar 14. PMID 36918157